CLINICAL TRIAL: NCT05069350
Title: A Double Blinded Randomized Controlled Study of Topical Anaesthetics Oxybuprocaine Versus Bupivacaine 0.5% in Intravitreal Injections
Brief Title: Bupivacaine vs Oxybuprocaine Topical Anesthesia in IVI
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Research Institute of Ophthalmology, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Topical anesthesia in IVI
Record Dates: First submitted 2021-09-14; First posted 2021-10-06 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: double blinded randomized syudy
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bupivacaine 0.5% (Experimental)
  Interventions: Drug: bupivacaine 0.5% and oxubuprocaine
- oxybuprocaine (Experimental)
  Interventions: Drug: bupivacaine 0.5% and oxubuprocaine

INTERVENTIONS:
Drug: bupivacaine 0.5% and oxubuprocaine — using each drug as surface anesthesia before intravitreal injections

SUMMARY:
comparing two local anaesthetic agents, Bupivacaine 0.5% versus Oxybuprocaine used topically to provide surface anaesthesia before IVI procedures.

DETAILED DESCRIPTION:
In preparation zone, we will cannulate the patients, connect them to the pulse oximetry and we will start providing appropriate surface anaesthesia for an adequate period of time before the patient administration of the injection, by applying the anaesthetic agents, 3 times with 5 minutes interval, for 15 minutes and then waitng the injection

All patients are informed that they are going to receive topical anaesthetic agent before the IVI.

pain is monitored during the injection by using the 11 points verbal numerical pain scaling as zero is for no pain and 10 is for severe unbearable pain.

ELIGIBILITY:
Inclusion Criteria:

* All patients between 30 to 70 years

Exclusion Criteria:

* uncooperative patients

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
verbal pain numerical scaling | 10 minutes
  11 point scale from 0-10 zero measns No pain 10 means severe unbearable pain

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Ophthamology, Giza, Haram, Egypt

IPD SHARING:
Plan to Share IPD: No